CLINICAL TRIAL: NCT07198451
Title: Efficacy Evaluation of Submucosal Injection of Gemcitabine in Preventing Recurrence of Intermediate- and High-Risk Non-Muscle-Invasive Bladder Cancer: A Randomized, Single-Blind, Multicenter Clinical Study
Brief Title: Efficacy of Gemcitabine Submucosal Injection for Preventing Recurrence in Intermediate- and High-Risk Non-Muscle-Invasive Bladder Cancer: A Randomized Trial
Acronym: GEM-IR-NMIBC
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Naiwen Chen, Resident physicians, Shanghai University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-1871-211-01
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Non Muscle Invasive Bladder Cancer
Keywords: non muscle invasive bladder cancer; Gemcitabine; Submucosal Injection; Recurrence; Randomized Controlled Trial
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Recurrence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gemcitabine Submucosal Injection Arm (Experimental): Patients in this arm will receive submucosal injections of gemcitabine following transurethral resection of bladder tumor (TURBT). The regimen consists of one injection immediately after TURBT, followed by additional injections once every three months, for a total of four injections. Each injection uses 1000mg of gemcitabine. Injection sites are planned based on bladder area and common tumor locations, administered using a specialized injection gun.
  Interventions: Drug: Gemcitabine Submucosal Injection
- Gemcitabine Intravesical Instillation Arm (Active Comparator): Patients in this arm will receive standard intravesical instillation of gemcitabine following TURBT. The regimen consists of one instillation immediately after surgery, followed by an induction phase of once-weekly instillations for eight weeks, and then a maintenance phase of once-monthly instillations for ten months. Each instillation uses 2000mg of gemcitabine dissolved in 50mL of normal saline, retained for 30-60 minutes.
  Interventions: Drug: Gemcitabine Intravesical Instillation

INTERVENTIONS:
Drug: Gemcitabine Submucosal Injection — A chemotherapeutic agent. Administered via submucosal injection into the bladder wall using a specialized injection gun. Dosage: 1000mg per injection. Regimen: One injection immediately post-TURBT, followed by one injection every three months for a total of four injections.
  Arms: Gemcitabine Submucosal Injection Arm
Drug: Gemcitabine Intravesical Instillation — Standard therapy. Administered by instilling a solution into the bladder via a catheter. Dosage: 2000mg dissolved in 50mL normal saline per instillation. Regimen: One instillation immediately post-TURBT, followed by an induction phase (once weekly for 8 weeks) and a maintenance phase (once monthly for 10 months). The solution is retained for 30-60 minutes.
  Arms: Gemcitabine Intravesical Instillation Arm

SUMMARY:
Bladder cancer is the most common malignant tumor of the urinary system in China, and its incidence has been increasing year by year. It is classified into non-muscle-invasive bladder cancer (NMIBC) and muscle-invasive bladder cancer (MIBC). NMIBC accounts for 75% of newly diagnosed bladder cancer cases, and transurethral resection of bladder tumor (TURBT) followed by postoperative intravesical therapy is the standard treatment for NMIBC. However, the 5-year recurrence rate of NMIBC remains as high as 50%, with 20-30% of patients progressing to MIBC. MIBC is characterized by rapid progression and a high tendency for metastasis. The 5-year survival rate for patients with metastatic bladder cancer is only 5.4%. This study aims to investigate the efficacy of submucosal injection of the chemotherapeutic agent gemcitabine in preventing recurrence of intermediate- and high-risk NMIBC. Additionally, it seeks to develop software and devices related to submucosal injection to promote the clinical application of this new approach in the chemotherapeutic management of NMIBC. This research is expected to bring a revolutionary breakthrough in the standardisation of whole-process diagnosis and treatment of NMIBC, holding significant scientific value and major clinical translational importance for improving therapeutic outcomes and prognosis of bladder cancer.

DETAILED DESCRIPTION:
Bladder cancer is a common malignant tumor of the urinary system. Globally, in 2023, there were approximately 610,000 new cases of bladder cancer and about 220,000 deaths attributed to the disease. In China, over the past two decades, the age-standardized incidence and prevalence rates of bladder cancer in men have increased by 71.79% and 195.38%, respectively. Over the last 15 years, the average annual mortality rate for male bladder cancer has risen by 3.84%, posing a serious threat to public health.

Bladder cancer is classified into non-muscle-invasive bladder cancer (NMIBC) and muscle-invasive bladder cancer (MIBC) based on whether the tumor invades the muscle layer. NMIBC accounts for approximately 75% of newly diagnosed bladder cancer cases. The standard treatment for NMIBC involves transurethral resection of bladder tumor (TURBT) followed by postoperative intravesical therapy. However, NMIBC often recurs within one year, with a recurrence rate as high as 60-70%, and 20-30% of cases progress to MIBC. Once bladder cancer advances to MIBC, it is characterized by rapid progression and a high tendency for metastasis. The standard treatment for MIBC is radical cystectomy with lymph node dissection, often accompanied by neoadjuvant or adjuvant chemotherapy. Traditional radical surgery for bladder cancer is highly invasive, associated with slow postoperative recovery and a high incidence of complications. The objective response rate for neoadjuvant or adjuvant chemotherapy is less than 50%. The 5-year survival rate for MIBC is below 60%, and for patients with distant metastasis, it drops significantly to just 5.4%.

In recent years, cancer immunotherapy, particularly immune checkpoint inhibitors, has advanced rapidly. However, immunotherapy also suffers from a low objective response rate, which is even below 30% in MIBC. Therefore, the high incidence, recurrence rate, and difficulty in curing bladder cancer remain significant challenges for both clinicians and patients.

TURBT is the standard surgical procedure for NMIBC. Intravesical therapy is a local adjuvant treatment used after TURBT to prevent recurrence. However, the efficacy of intravesical therapy is limited by inadequate drug absorption, resulting in insufficient local drug concentrations and suboptimal therapeutic outcomes. Moreover, postoperative intravesical therapy involves long-term, repeated invasive procedures, which often lead to complications such as urinary tract infections, bladder irritation, and urethral strictures. Improving the efficiency of drug utilization in intravesical therapy is a promising approach to address these issues. Enhancing drug absorption and prolonging the sustained-release effect of the agents could improve treatment efficacy while reducing the frequency of intravesical instillations, ultimately improving the prognosis of NMIBC, lowering recurrence rates, and reducing the risk of progression to MIBC. Submucosal injection of chemotherapeutic drugs offers a potential solution by increasing drug utilization efficiency and reducing complications associated with intravesical therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 80 years (inclusive) with radiologically confirmed bladder tumor and scheduled to undergo transurethral resection of bladder tumor (TURBT).
2. Postoperative pathological confirmation of intermediate- or high-risk non-muscle-invasive bladder cancer (NMIBC).
3. Voluntarily participate in the study and sign the informed consent form, ensuring the patient fully understands the trial purpose, risks, and right to withdraw.

Exclusion Criteria:

1. Preoperative comorbidities including detrusor overactivity, urethral stricture, urge incontinence, stress incontinence, or overflow incontinence.
2. Concurrent urogenital infectious diseases (e.g., acute urethritis, acute cystitis).
3. History of pelvic radiotherapy.
4. Receiving systemic anti-tumor therapy for any malignant tumor.
5. Severe cardiovascular disease, hepatic or renal insufficiency, or coagulation dysfunction.
6. Presence of mental illness or psychological disorders that impair normal communication.
7. Any other situation deemed by the investigator as unsuitable for participation in this clinical study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
24-month Bladder Tumor Recurrence Rate | 24 months post-operation
  The proportion of patients with bladder tumor recurrence confirmed by cystoscopy and tissue biopsy within 24 months after transurethral resection of bladder tumor (TURBT). The recurrence rate is calculated as: (Number of patients with confirmed recurrence in the group / Total number of analyzed patients in that group) × 100%.

SECONDARY OUTCOMES:
Proportion of Pathological Grade Upgrading upon Recurrence | Through study completion, up to 60 months
  The proportion of patients with recurrent tumor whose pathological grade (e.g., from low-grade to high-grade) is worse than at initial diagnosis among all patients with recurrence.
Tumor Complete Response (CR) Rate | Through study completion, up to 60 months
  The proportion of patients with no evidence of tumor recurrence, metastasis, or progression as confirmed by regular cystoscopy, biopsy, urinary cytology, and imaging.
Incidence of Bladder Irritation Symptoms and Gross Hematuria | Through study completion, up to 60 months
  Record and compare the proportion of patients in both groups experiencing bladder irritation symptoms (e.g., frequency, urgency, dysuria) and gross hematuria post-operation.
Change in Quality of Life Core Questionnaire (QLQ-C30) Score | Through study completion, up to 60 months
  Assessed using the EORTC QLQ-C30 questionnaire. It includes 5 functional scales, 3 symptom scales, and a global health status item. The change from baseline in scores will be used to evaluate the change in quality of life.
Change in Bladder Cancer-Specific Module (QLQ-BLM30) Score | Through study completion, up to 60 months
  Assessed using the EORTC QLQ-BLM30 module. It evaluates bladder cancer-specific quality of life dimensions such as urinary symptoms, physical function, and psychological state. The change from baseline in scores will be used for evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Dongliang Xu, Principal Investigator — Shuguang Hospital Affiliated to Shanghai University of Traditional Chinese Medicine

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in the primary publications of this trial will be shared. This includes data on demographics, tumor characteristics, treatment allocation, recurrence, progression, safety, and quality of life scores.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD and supporting documents will become available following the publication of the primary results in a peer-reviewed journal. There is no end date for data sharing.
Access Criteria: Data will be accessible to researchers who provide a methodologically sound proposal for approved purposes. Proposals should be directed to the corresponding author. Requestors will need to sign a data access agreement to gain access. A committee led by the principal investigator will review proposals.

REFERENCES:
- [Background] Liu K, Peng J, Guo Y, Li Y, Qi X, Duan D, Li T, Li J, Niu Y, Han G, Zhao Y. Expanding the Potential of Neoantigen Vaccines: Harnessing Bacille Calmette-Guerin Cell-Wall-Based Nanoscale Adjuvants for Enhanced Cancer Immunotherapy. ACS Nano. 2024 May 7;18(18):11910-11920. doi: 10.1021/acsnano.4c01691. Epub 2024 Apr 29. PMID 38680054
- [Background] Koya MP, Simon MA, Soloway MS. Complications of intravesical therapy for urothelial cancer of the bladder. J Urol. 2006 Jun;175(6):2004-10. doi: 10.1016/S0022-5347(06)00264-3. PMID 16697786
- [Background] Gravestock P, Cullum D, Somani B, Veeratterapillay R. Diagnosing upper tract urothelial carcinoma: A review of the role of diagnostic ureteroscopy and novel developments over last two decades. Asian J Urol. 2024 Apr;11(2):242-252. doi: 10.1016/j.ajur.2022.08.003. Epub 2022 Sep 23. PMID 38680592
- [Background] Morad G, Helmink BA, Sharma P, Wargo JA. Hallmarks of response, resistance, and toxicity to immune checkpoint blockade. Cell. 2021 Oct 14;184(21):5309-5337. doi: 10.1016/j.cell.2021.09.020. Epub 2021 Oct 7. PMID 34624224
- [Background] Kartolo A, Robinson A, Vera Badillo FE. Can Oncogenic Driver Alterations be Responsible for the Lack of Immunotherapy Efficacy in First-line Advanced Urothelial Carcinoma? Eur Urol. 2023 Jan;83(1):1-2. doi: 10.1016/j.eururo.2022.04.022. Epub 2022 May 20. PMID 35606230
- [Background] Powles T, Park SH, Voog E, Caserta C, Valderrama BP, Gurney H, Kalofonos H, Radulovic S, Demey W, Ullen A, Loriot Y, Sridhar SS, Tsuchiya N, Kopyltsov E, Sternberg CN, Bellmunt J, Aragon-Ching JB, Petrylak DP, Laliberte R, Wang J, Huang B, Davis C, Fowst C, Costa N, Blake-Haskins JA, di Pietro A, Grivas P. Avelumab Maintenance Therapy for Advanced or Metastatic Urothelial Carcinoma. N Engl J Med. 2020 Sep 24;383(13):1218-1230. doi: 10.1056/NEJMoa2002788. Epub 2020 Sep 18. PMID 32945632
- [Background] Advanced Bladder Cancer (ABC) Meta-analysis Collaborators Group. Adjuvant Chemotherapy for Muscle-invasive Bladder Cancer: A Systematic Review and Meta-analysis of Individual Participant Data from Randomised Controlled Trials. Eur Urol. 2022 Jan;81(1):50-61. doi: 10.1016/j.eururo.2021.09.028. Epub 2021 Nov 19. PMID 34802798
- [Background] Cambier S, Sylvester RJ, Collette L, Gontero P, Brausi MA, van Andel G, Kirkels WJ, Silva FC, Oosterlinck W, Prescott S, Kirkali Z, Powell PH, de Reijke TM, Turkeri L, Collette S, Oddens J. EORTC Nomograms and Risk Groups for Predicting Recurrence, Progression, and Disease-specific and Overall Survival in Non-Muscle-invasive Stage Ta-T1 Urothelial Bladder Cancer Patients Treated with 1-3 Years of Maintenance Bacillus Calmette-Guerin. Eur Urol. 2016 Jan;69(1):60-9. doi: 10.1016/j.eururo.2015.06.045. Epub 2015 Jul 23. PMID 26210894
- [Background] Comperat E, Amin MB, Cathomas R, Choudhury A, De Santis M, Kamat A, Stenzl A, Thoeny HC, Witjes JA. Current best practice for bladder cancer: a narrative review of diagnostics and treatments. Lancet. 2022 Nov 12;400(10364):1712-1721. doi: 10.1016/S0140-6736(22)01188-6. Epub 2022 Sep 26. PMID 36174585
- [Background] Lopez-Beltran A, Cookson MS, Guercio BJ, Cheng L. Advances in diagnosis and treatment of bladder cancer. BMJ. 2024 Feb 12;384:e076743. doi: 10.1136/bmj-2023-076743. PMID 38346808
- [Background] Qi J, Li M, Wang L, Hu Y, Liu W, Long Z, Zhou Z, Yin P, Zhou M. National and subnational trends in cancer burden in China, 2005-20: an analysis of national mortality surveillance data. Lancet Public Health. 2023 Dec;8(12):e943-e955. doi: 10.1016/S2468-2667(23)00211-6. PMID 38000889
- [Background] Bray F, Laversanne M, Sung H, Ferlay J, Siegel RL, Soerjomataram I, Jemal A. Global cancer statistics 2022: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2024 May-Jun;74(3):229-263. doi: 10.3322/caac.21834. Epub 2024 Apr 4. PMID 38572751